CLINICAL TRIAL: NCT02876172
Title: A Phase 1/2 Open-Label Treatment Development Study of Methylenedioxymethamphetamine (MDMA)-Assisted Cognitive-Behavioral Conjoint Therapy (CBCT) in Dyads in Which 1 Member Has Chronic Posttraumatic Stress Disorder (PTSD)
Brief Title: MDMA-Assisted Cognitive-Behavioral Conjoint Therapy (CBCT) in Dyads in Which 1 Member Has Chronic PTSD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPVA-1
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; therapy; MDMA; dyad; cognitive behavioral therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDMA-assisted therapy and CBCT (Experimental): Cognitive-behavioral conjoint therapy and 2 sessions of MDMA-assisted therapy.
  Interventions: Drug: MDMA; Behavioral: CBCT; Behavioral: Therapy

INTERVENTIONS:
Drug: MDMA — Two sessions of MDMA-assisted therapy, one with an initial dose of 75 mg midomafetamine HCl (and optional supplemental dose of 37.5 mg) and the second with 75 or 100 mg midomafetamine HCl (with optional supplemental dose of either 37.5 mg or 50 mg respectively) given to the participant with PTSD and their significant other.
  Other Names: 3,4-Methylenedioxymethamphetamine; midomafetamine
Behavioral: CBCT — A three-phase, 15-session, manualized treatment from the CBCT manual
  Other Names: Cognitive behavioral conjoint therapy
Behavioral: Therapy — Manualized MDMA-assisted therapy

SUMMARY:
The goal of this clinical trial is to learn if cognitive-behavioral conjoint therapy (CBCT) in combination with MDMA-assisted therapy is safe and effective in people with chronic PTSD and their partners.

The main question it aims to answer is: Does MDMA-assisted CBCT reduce PTSD symptoms in people with chronic PTSD?

Participants (chronic PTSD patients and their partners) will undergo three non-drug preparatory therapy sessions, followed by two MDMA-assisted therapy sessions. Each MDMA-assisted therapy session will be followed by five non-drug integrative therapy using CBCT.

DETAILED DESCRIPTION:
Cognitive-Behavioral Conjoint Therapy (CBCT) for PTSD is a three-phase, 15-session, manualized treatment. This Phase 1/2 open-label study will combine methods for conducting MDMA-assisted therapy with methods from the CBCT for PTSD in order to treat 10 participants with chronic PTSD and their partners (intimate or non-intimate significant other who does not have a current diagnosis of PTSD) in order to explore whether combined treatment is effective.

Each therapy team will have one therapist trained and experienced in MDMA-assisted therapy and one therapist trained and experienced in CBCT. During the first experimental session, both participants will receive 75 mg of midomafetamine HCl followed 1.5 to 2 hours later by an optional supplemental half-dose of 37.5 mg. During the second experimental session, an initial dose of either 100 or 75 mg of midomafetamine HCl will be administered to both participants followed by an optional supplemental half-dose of either 50 mg or 37.5 mg. The primary objective of this study is to assess changes in PTSD symptoms from Baseline to Primary Endpoint in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total severity scores in PTSD participants.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria for the PTSD and Concerned Significant Other (CSO) are identical except for first two items, marked below:
* PTSD+ participant: Meet DSM-5 criteria for current PTSD and satisfies PTSD criteria via CAPS
* CSO participant: Meet criteria for V62.89 Other Problem Related to Psychosocial Circumstances under Diagnostic and Statistical Manual 5 (DSM-5), as determined through clinical interview, for current psychosocial circumstances contributing to relationship distress with intimate or non-intimate partner
* Are at least 18 years old
* If in psychotherapy, willing and able to maintain that schedule without changing it
* Are willing to refrain from taking any psychiatric medications during the study period, with the exception of gabapentin when prescribed for pain control.
* Willing to remain overnight at the study site
* Are willing to be driven home the morning after the experimental sessions, after the integrative therapy session
* Are willing to commit to medication dosing, experimental sessions, follow-up sessions, to complete evaluation instruments and commit to be contacted for all necessary telephone contacts
* Are willing to remain overnight at the study site after each experimental session until after the integrative session occurring the next morning
* Must have a negative pregnancy test at study entry and prior to each experimental session if able to bear children, and must agree to use adequate birth control through 10 days after the last dose of MDMA.
* Must provide a contact (relative, spouse, close friend or other caregiver other than the CSO participant) who is willing and able to be reached by the Clinical Investigators in the event of a participant becoming suicidal.
* Must agree to inform the Clinical Investigators within 48 hours of any medical conditions and procedures
* Are proficient in speaking and reading English
* Agree to have all clinic visit and Integrative Sessions recorded to audio and video
* Agree to not participate in any other interventional clinical trials during the duration of this study

Exclusion Criteria:

* The following exclusions are identical for PTSD+ and CSO participants except for the following, marked below:
* CSO participant only: Have diagnosis of current PTSD not in remission
* Are pregnant or nursing, or are women of child bearing potential who are not practicing an effective means of birth control
* Have evidence or history of significant medical disorders
* Have hypertension
* Have liver disease; asymptomatic participants with Hepatitis C who have previously undergone evaluation and successful treatment is permitted.
* History of hyponatremia or hyperthermia
* Weigh less than 48 kg
* Have used "Ecstasy" (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the MDMA-assisted session
* Are not able to give adequate informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-03 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Mithoefer, MD, Principal Investigator — Private Practice
Locations (1):
- Offices of Michael Mithoefer MD, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share outcome measure data upon request
Supporting Information: Study Protocol, SAP
Time Frame: After study data lock

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient MDMA and CBCT; Partner MDMA and CBCT: Cognitive-behavioral conjoint therapy and 2 sessions of MDMA-assisted psychotherapy.
  MDMA: Two sessions of MDMA-assisted psychotherapy, one with an initial dose of 75 mg (and optional supplemental dose of 37.5 mg) and the second with 75 or 100 mg MDMA (with optional supplemental dose of either 37.5 mg or 50 mg respectively) given to the participant with PTSD and their significant other.
  CBCT: A three-phase, 15-session, manualized treatment from the CBCT manual
  Therapy: Non-directive therapy (from MAPS MDMA-assisted therapy treatment manual)
Period: Overall Study
Arm/Group | Patient MDMA and CBCT | Partner MDMA and CBCT
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient MDMA and CBCT | Partner MDMA and CBCT | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.54) | 46.5 (11.17) | 46.8 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Global CAPS-5 Total Severity Score [Mean (Standard Deviation); unit: units on a scale] — Population: Partner does not have PTSD therefore CAPS-5 was not assessed per protocol
  units on a scale
    number analyzed (Participants) | 6 | 0 | 6
    (all) | 42.0 (5.76) |  | 42.0 (5.76)

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a CAPS-5 total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MDMA (75 mg or 100 mg) + CBCT: Cognitive-behavioral conjoint therapy and 2 sessions of MDMA-assisted psychotherapy.
  MDMA: Two sessions of MDMA-assisted psychotherapy, one with an initial dose of 75 mg (and optional supplemental dose of 37.5 mg) and the second with 75 or 100 mg MDMA (with optional supplemental dose of either 37.5 mg or 50 mg respectively) given to the participant with PTSD and their significant other.
  CBCT: A three-phase, 15-session, manualized treatment from the CBCT manual
  Therapy: Non-directive therapy (from MAPS MDMA-assisted therapy treatment manual)
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 16.3 (13.71)

2. Primary Outcome: Change From Baseline to Primary Endpoint CAPS-5 Total Severity Score
Description: as for outcome 1
Time Frame: Baseline to Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD Patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | -25.7 (13.89)

3. Secondary Outcome: Baseline Pittsburgh Sleep Quality Index (PSQI)
Description: Self-reported questionnaire that assesses sleep quality and disturbances. The index looks at subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The component scores yield a total score which ranges 0-21 with a higher score indicating worse sleep quality.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 14.24 (3.54)

4. Secondary Outcome: Primary Endpoint Pittsburgh Sleep Quality Index (PSQI)
Description: as for outcome 3
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 10.37 (4.49)

5. Secondary Outcome: Baseline Patient Beck Depression Inventory-II (BDI-II)
Description: BDI-II is a 21-item self reported instrument used to measure severity of depressive symptoms. The BDI-II total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depressive symptoms. The scores range from 0 to 63, with higher score indicating greater severity of depressive symptoms.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 32.91 (8.75)

6. Secondary Outcome: Primary Endpoint Patient Beck Depression Inventory-II (BDI-II)
Description: as for outcome 5
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 12.75 (16.88)

7. Secondary Outcome: Baseline Patient Couples Satisfaction Index (CSI)
Description: The Couples Satisfaction Index (CSI) is a self-reported 32-item scale measuring one's satisfaction in a relationship. Questions discuss overall happiness in relationship, extent of agreement/ disagreement between partners, and feelings towards relationships and are scored on a likert scale from 0 to 5, with higher scores indicating higher satisfaction in the relationship. Scores range from 0 to 160.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 105.37 (13.39)

8. Secondary Outcome: Primary Endpoint Patient Couples Satisfaction Index (CSI)
Description: as for outcome 7
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 127.00 (34.34)

9. Secondary Outcome: Baseline Partner Couples Satisfaction Index (CSI)
Description: as for outcome 7
Time Frame: Baseline (screening)
Population: PTSD patient's partner
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 98.1 (50.81)

10. Secondary Outcome: Primary Endpoint Partner Couples Satisfaction Index (CSI)
Description: as for outcome 7
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient's partner
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 125.34 (30.59)

11. Secondary Outcome: Baseline Trauma and Attachment Beliefs Scale (TABS)
Description: TABS is a 84-item self-report scale, which measures responses on a 1 to 6 scale (1 = "Disagree Strongly, 6 = Agree Strongly) the degree to which respondents believe the statements correspond with their own beliefs. The measures of these beliefs relate to self-safety, other-safety, self-trust, other-trust, self-esteem, other-esteem, self-intimacy, other-intimacy, self-control, and other control. A TABS total score is calculated by summing all of the items (range 84 to 504). Higher scores indicate greater disruption.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 289.78 (44.30)

12. Secondary Outcome: Primary Endpoint Trauma and Attachment Beliefs Scale (TABS)
Description: as for outcome 11
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 232.7 (69.07)

13. Secondary Outcome: Baseline Emotion Regulation Questionnaire (ERQ) Reappraisal Subscale
Description: ERQ measures self-reported emotional regulation and includes 10 items to assess means of coping with emotions via regulating them through reappraisal or suppression. Items range from 1 (strongly disagree) to 7 (strongly agree). Six of the items are summed to create the reappraisal total score, with total scores ranging from 6 to 42. Higher scores indicate greater emotional reappraisal.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 21.77 (7.92)

14. Secondary Outcome: Primary Endpoint Emotion Regulation Questionnaire (ERQ) Reappraisal Subscale
Description: as for outcome 13
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 28.34 (2.30)

15. Secondary Outcome: Baseline Emotion Regulation Questionnaire (ERQ) Suppression Subscale
Description: ERQ measures self-reported emotional regulation and includes 10 items to assess means of coping with emotions via regulating them through reappraisal or suppression. Items range from 1 (strongly disagree) to 7 (strongly agree). Four of the items are summed to create the suppression total score, with total scores ranging from 4 to 28. Higher scores indicate greater emotional suppression.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 18.96 (6.28)

16. Secondary Outcome: Primary Endpoint Emotion Regulation Questionnaire (ERQ) Suppression Subscale
Description: as for outcome 15
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 13.63 (5.41)

17. Secondary Outcome: Baseline Patient PTSD Checklist-5 (PCL-5)
Description: The PTSD Checklist-5 (PCL-5) is a 20-item self-reported questionnaire that follows DSM-5 criteria to assess PTSD presence and severity. Item scores range from 0 (not at all) to 4 (extremely). A total symptom severity score is determined by summing all items (range 0 to 80). A higher score indicates greater PTSD symptom severity.
Time Frame: Baseline (screening)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 62.64 (6.35)

18. Secondary Outcome: Primary Endpoint Patient PTSD Checklist-5 (PCL-5)
Description: as for outcome 17
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 23.96 (19.08)

19. Secondary Outcome: Baseline Partner-rated PTSD Checklist-5 (PCL-5)
Description: as for outcome 17
Time Frame: Baseline (screening)
Population: PTSD patient's partner
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 49.58 (8.52)

20. Secondary Outcome: Primary Endpoint Partner-rated PTSD Checklist-5 (PCL-5)
Description: as for outcome 17
Time Frame: Primary Endpoint (Visit 16, approximately 2 months later)
Population: PTSD patient's partner
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA (75 mg or 100 mg) + CBCT
Number analyzed (Participants) | 6
score on a scale | 21.54 (19.67)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to study completion (a period of approximately 6 months) and at 6-month follow-up (1 year after enrollment).
Groups:
- PTSD Patients Open-label CBCT and MDMA-assisted Therapy (up to 2 Months Post Last Experimental Dose); CSO Patients Open-label CBCT and MDMA-assisted Therapy (up to 2 Months Post Last Experimental Dose); PTSD Patients at 6-month Follow-up; CSO Patients at 6-month Follow-up: Cognitive-behavioral conjoint therapy and 2 sessions of MDMA-assisted therapy.
  MDMA: Two sessions of MDMA-assisted psychotherapy, one with an initial dose of 75 mg (and optional supplemental dose of 37.5 mg) and the second with 75 or 100 mg MDMA (with optional supplemental dose of either 37.5 mg or 50 mg respectively) given to the participant with PTSD and their significant other.
  CBCT: A three-phase, 15-session, manualized treatment from the CBCT manual
  Therapy: Non-directive therapy (from MAPS MDMA-assisted therapy treatment manual)
Arm/Group | PTSD Patients Open-label CBCT and MDMA-assisted Therapy (up to 2 Months Post Last Experimental Dose) | CSO Patients Open-label CBCT and MDMA-assisted Therapy (up to 2 Months Post Last Experimental Dose) | PTSD Patients at 6-month Follow-up | CSO Patients at 6-month Follow-up
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PTSD Patients Open-label CBCT and MDMA-assisted Therapy (up to 2 Months Post Last Experimental Dose) (N=6) | CSO Patients Open-label CBCT and MDMA-assisted Therapy (up to 2 Months Post Last Experimental Dose) (N=6) | PTSD Patients at 6-month Follow-up (N=6) | CSO Patients at 6-month Follow-up (N=6)
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion, spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Tic (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT02876172/Prot_003.pdf
  • Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02876172/SAP_001.pdf
  • Informed Consent Form (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT02876172/ICF_002.pdf